CLINICAL TRIAL: NCT00757848
Title: A Phase II, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy of 28 Day Oral Administration of AZD9668 in Patients With Cystic Fibrosis
Brief Title: A Phase II , Placebo-controlled Study to Assess Efficacy of 28 Day Oral AZD9668 in Patients With Cystic Fibrosis
Acronym: INCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0520C00009
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD9668 (Experimental)
  Interventions: Drug: AZD9668
- Placebo (Placebo Comparator)
  Interventions: Drug: AZD9668 Placebo equivalent

INTERVENTIONS:
Drug: AZD9668 — 60 mg, oral tablet, twice daily for 28 days
  Arms: AZD9668
Drug: AZD9668 Placebo equivalent — Match placebo to 60 mg, oral tablet, twice daily for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate if treatment with AZD9668 for 28 days is effective in treating Cystic Fibrosis (CF) and if so how it compares to placebo (a substance which does not have any action).

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal or surgically sterile female patients
* Have a clinical diagnosis of Cystic Fibrosis with lung function tests greater or equal to 40% of normal
* Have normal renal function

Exclusion Criteria:

* Lung transplant patients
* Significant liver disease
* Any other non-CF-related lung disease that may interfere with study assessments

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Elborn, Principal Investigator — Belfast hospital; Joanna Marks-Konczalik, Study Director — AstraZeneca
Locations (14):
- Research Site, Copenhagen, Denmark
- Germany (4):
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, München
- Poland (2):
  - Research Site, Rabka-Zdrój
  - Research Site, Warsaw
- Research Site, Moscow, Russia
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala
- United Kingdom (2):
  - Research Site, Belfast, Northern Ireland
  - Research Site, Liverpool

REFERENCES:
- [Derived] Elborn JS, Perrett J, Forsman-Semb K, Marks-Konczalik J, Gunawardena K, Entwistle N. Efficacy, safety and effect on biomarkers of AZD9668 in cystic fibrosis. Eur Respir J. 2012 Oct;40(4):969-76. doi: 10.1183/09031936.00194611. Epub 2012 Jan 20. PMID 22267768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 30 October 2008. Last patient completed 04 August 2009. Study conducted at 15 centres in 6 countries (UK, Germany, Sweden, Poland, Denmark, Russia).
Groups:
- AZD9668: AZD9668, 2 x 30 mg twice daily (bid)
- Placebo: Placebo, 2 tablets twice daily (bid)
Period: Overall Study
Arm/Group | AZD9668 | Placebo
Started | 27 | 29
Completed | 24 | 27
Not Completed | 3 | 2
Not completed — Voluntary discontinuation | 1 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Incorrect enrolment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9668 | Placebo | Total
Number analyzed (Participants) | 25 | 29 | 54
Age Continuous [Median (Full Range); unit: years] | 25 [20 to 51] | 25 [17 to 53] | 25 [17 to 53]
Sex: Female, Male [Count of Participants; unit: Participants] — Two patients excluded from analysis set. No data for patient who prematurely discontinued and for patient who did not receive any study medication.
  Participants
    Female | 1 | 0 | 1
    Male | 24 | 29 | 53

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Sputum Absolute Neutrophil Count at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: Baseline and Values from day 21 to 28
Population: The efficacy analysis set for each outcome measure includes those patients who received at least one dose of investigational product and for whom a baseline and at least one post-randomisation measurement is available for that outcome measure. Patients were analysed by to randomised treatment in accordance with the intention to treat principle.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 1.07 [0.82 to 1.40] | 1.10 [0.86 to 1.41]

2. Primary Outcome: Sputum Percentage Neutrophil Count
Description: Percentage of neutrophils in white blood cell count.Change from Baseline (mean of 2 baseline visits) to the end of the treatment period (mean of 2 visits at the end of the treatment)
Time Frame: Baseline and Values from day 21 to 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of neutrophils in WBCs
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
percentage of neutrophils in WBCs | 3.21 (1.757) [lower limit 1.757] | 1.96 (1.566) [lower limit 1.566]

3. Primary Outcome: 24-hour Sputum Weight
Description: Sputum weight (g) collected during 24 hour periods. Change from Baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 27
grams | -2.29 (2.261) [lower limit 2.261] | -5.13 (2.178) [lower limit 2.178]

4. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function.Change from Baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 29
L | -0.02 (0.048) [lower limit 0.048] | 0.01 (0.043) [lower limit 0.043]

5. Primary Outcome: Slow Vital Capacity (SVC)
Description: Slow Vital capacity (L) as a measure of lung function. Change from Baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 27
L | -0.03 (0.106) [lower limit 0.106] | -0.15 (0.081) [lower limit 0.081]

6. Primary Outcome: Forced Expiratory Flow Between 25 and 75% of Forced Vital Capacity (FEF25-75%)
Description: FEF25-75% (L) as a measure of lung function. Change from Baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 29
L | -0.07 (0.090) [lower limit 0.090] | 0.08 (0.082) [lower limit 0.082]

7. Primary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (L) as a measure of lung function. Change from Baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 29
L | -0.06 (0.066) [lower limit 0.066] | 0.01 (0.059) [lower limit 0.059]

8. Primary Outcome: Morning Peak Expiratory Flow (PEF)
Description: Morning Peak Expiratory Flow (L/min) as a measure of lung function.Change from baseline value to mean of the last 7 days on treatment
Time Frame: Last 7 days on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 29
L/min | -1.17 (8.055) [lower limit 8.055] | 14.05 (7.262) [lower limit 7.262]

9. Primary Outcome: Evening Peak Expiratory Flow (PEF)
Description: Evening Peak Expiratory Flow (L/min) as a measure of lung function.Change from baseline value to mean of the last 7 days on treatment
Time Frame: The last 7 days on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 29
L/min | 0.59 (6.874) [lower limit 6.874] | 6.32 (6.194) [lower limit 6.194]

10. Primary Outcome: Bronkotest Diary Card Signs and Symptoms
Description: The Bronkotest diary card includes 8 questions on signs and symptoms. Symptom scores were recorded for night-time symptoms, breathing, sputum colour, sputum amount, sputum type, wellbeing, and cough, generally scored on a scale from 0 (no symptoms) to 4 (worst symptoms). ANOVA models were fitted to compare the change from baseline between AZD9668 and placebo for each question separately, with a p-value of 0.1 considered statistically significant. The number of number of these 8 measures with significant differences is reported.
Time Frame: The last 7 days on treatment
Population: as for outcome 1
Measure: Number; unit: Signs and Symptoms
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 29
Signs and Symptoms | 0 | 0

11. Primary Outcome: Cystic Fibrosis Questionnaire (CFQ-R) - Quittner
Description: Cystic Fibrosis Questionnaire Overall Score as a measure of quality of life and disease symptoms. Scores range from 0 to 100, with higher scores indicating better health. The overall score is the sum of 12 subscores. Change from baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 27
units on a scale | -19.7 (18.12) [lower limit 18.12] | 4.7 (14.93) [lower limit 14.93]

12. Secondary Outcome: Ratio of Sputum Tumour Necrosis Factor Alpha (TNF α) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits.Values from day 21 to 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 0.91 [0.69 to 1.20] | 1.24 [0.97 to 1.60]

13. Secondary Outcome: Ratio of Sputum Interleukin 6 (IL-6) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 0.71 [0.56 to 0.90] | 1.20 [0.96 to 1.48]

14. Secondary Outcome: Ratio of Sputum Interleukin 1 Beta (IL-1β) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 0.95 [0.75 to 1.22] | 1.09 [0.87 to 1.36]

15. Secondary Outcome: Ratio of Sputum Regulated on Activation, Normal T Cell Expressed and Secreted (RANTES) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 0.91 [0.74 to 1.12] | 1.18 [0.98 to 1.42]

16. Secondary Outcome: Ratio of Sputum Monocyte Chemoattractant Protein-1 (MCP-1) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 28
ratio | 0.73 [0.60 to 0.88] | 0.91 [0.76 to 1.08]

17. Secondary Outcome: Ratio of Sputum Interleukin 8 (IL-8) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 26
ratio | 0.86 [0.71 to 1.05] | 1.04 [0.86 to 1.26]

18. Secondary Outcome: Ratio of Sputum Leukotriene B4 (LTB4) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 2 visits at the end of the treatment period to the mean of 2 baseline visits
Time Frame: End of treatment values from 2 visits (day 21 to 28) and baseline values from 2 visits
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 24 | 25
ratio | 1.02 [0.87 to 1.19] | 1.00 [0.86 to 1.17]

19. Secondary Outcome: Ratio of Urine Desmosine (Free) (Normalised for Creatinine) at End of Treatment Compared to Baseline
Description: Ratio of day 28 to baseline
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 25
ratio | 0.88 [0.76 to 1.03] | 1.27 [1.08 to 1.48]

20. Secondary Outcome: Ratio of Urine Desmosine (Total) (Normalised for Creatinine) at End of Treatment Compared to Baseline
Description: Ratio of day 28 to baseline
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 22 | 27
ratio | 0.68 [0.53 to 0.87] | 0.97 [0.78 to 1.22]

ADVERSE EVENTS:
Description: Safety analysis set - one patient not included as he/she did not receive any study drug.
Arm/Group | AZD9668 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/29
Other Adverse Events (participants affected / at risk) | 16/26 | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9668 (N=26) | Placebo (N=29)
Pneumonia (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9668 (N=26) | Placebo (N=29)
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No